CLINICAL TRIAL: NCT07356635
Title: Investigating Cardiovascular Reactivity and Recovery of Young Adults During Grief-Recall, With Self-Affirmation as Potential Intervention
Brief Title: Cardiovascular Effects of Grieving
Acronym: SAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Kaiyuan Luo, Principal Investigator, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY008302
Record Dates: First submitted 2025-12-29; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Grief; Cardiovascular Health; Emotion
Keywords: grief; cardiovascular reactivity; cardiovascular health; heart rate variability; psychophysiology; self-affirmation; value-affirmation; stress; mourning

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either value-affirmation treatment or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grief-reducing intervention (Experimental): Participants will be randomly assigned to either a self-affirming task or a non-affirming neutral task prior to engaging in grief recall.
  Interventions: Behavioral: Value-affirmation
- Control group (No Intervention): Participants will be randomly assigned to either a self-affirming task or a non-affirming neutral task prior to engaging in grief recall. Participants in no-affirmation control group will be asked to rank their top 12 favorite jellybean flavors and write about the 3rd and 4th favorite flavor for 10 minutes. This control task has also been tested to propose same amount of workload without promoting participants' self-worth.

INTERVENTIONS:
Behavioral: Value-affirmation — Participants who are randomly assigned to the value-affirmation condition will be presented with 11 values and qualities to rank in order of importance from 1 to 11. Values presented including: being creative / artistic, government or politics, independence, learning and gaining knowledge, athletic ability, belonging to a group (such as your community, cultural group, or school club), music, career, spiritual or religious values, sense of humor.
  Participants will then be asked to write about their top-ranked value/quality and how it makes them feel good about themselves for 10 minutes.
  Other Names: self-affirmation
  Arms: Grief-reducing intervention

SUMMARY:
Self-affirmation (SA) theory proposes that people are motivated to maintain a positive self-image of being worthy, stable, and capable. Self-affirmation (SA) manipulations have been shown to effectively increase self-worth as well as reduce cardiovascular reactivity while enhancing cardiovascular recovery in response to stress. While SA is discussed as a way to alleviate grief, its effect on cardiovascular reactivity (CVR) and recovery to grief recall has yet to be studied within laboratory settings. This study proposes an experimental design to examine how an in-lab manipulation promoting self-affirmation can improve patients' cardiovascular responses during and after a grief recall procedure. The investigators hypothesized that grief severity (a continuous variable) interacts with condition (a categorical variable with two levels, i.e., SA intervention vs. control) to predict CV reactivity and recovery as outcomes.

Primary Objective 1: To investigate effects of self-affirmation intervention on cardiovascular responses among grieving participants during and after grief recall.

Secondary Objective 1: To investigate the relationship of grief severity with psychological stress.

DETAILED DESCRIPTION:
Background

Grief refers to individual's emotional response to real, perceived, and anticipated loss, and is known to induce various psychological symptoms such as depression and anxiety and physical symptoms such as nausea, tension, or fatigue. If a grief reaction is prolonged and left untreated, it could lead to prolonged grief disorder and affect individuals' daily lives. More severe consequences, such as heightened mortality rates, have been observed among bereaved populations, particularly in relation to accidental, violent, and alcohol-related causes, where excess mortality ranges from 50% to 150%. These effects are more pronounced during short durations of bereavement (<6 months) compared to longer periods and are greater among younger individuals.

Grief is a kind of psychological stress that induces the fight-or-flight response, activating the autonomic nervous system (ANS) and the hypothalamic-pituitary-adrenal (HPA) axis, and in turn, promoting the elevation in the sympathetic nervous system which result in heightened heart rate, blood pressure, blood glucose levels, etc. Specifically, studies have revealed grief's influence on cardiovascular system. Cardiovascular biomarkers affected by short- and long-term bereavement include heightened cortisol levels, dysregulated HPA axis, and more. Many of the effects are long-lasting and highly determined by length of bereavement. For example, a previous study revealed that early bereavement is associated with increased 24-hour heart rate and decreased heart rate variability, and the effect is persistent through 6 months into bereavement. Studies have also shown that immediate grief (grief in response to death of a closed one within 6 months) is correlated with heightened cardiovascular reactivity (CVR) and impaired cardiovascular recovery.

Investigating grief within a laboratory setting presents methodological challenges; however, the Grief Recall (GR) interview offers a standardized approach to eliciting bereavement-related stress. Developed by Dr. Mary-Frances O'Connor at the University of Arizona, GR is an adaptation of the Anger Recall and Separation Recall tasks and utilizes a semi-structured interview to induce grief as the primary stressor. Findings indicate that GR elicits significant increases in systolic blood pressure (SBP) and diastolic blood pressure (DBP) from a resting state, with grief severity predicting the magnitude of SBP elevation. The present study builds upon this work by employing a larger sample size and expanding cardiovascular measurements beyond blood pressure to include heart rate (HR), respiratory sinus arrhythmia (RSA), and cardiac output (CO) and total peripheral resistance (TPR). This approach aims to provide a more comprehensive assessment of cardiovascular responses to grief elicitation within a controlled experimental framework.

Self-affirmation (SA) theory proposes that people are motivated to maintain a positive self-image of being worthy, stable, and capable. The theory also states that when facing threats, people engaging in self-affirmation resist negative consequences by maintaining a self-competent image. Studies have revealed that self-affirmation manipulation targets brain regions responsible for self-processing (medial prefrontal cortex and posterior cingulate cortex), as well as valuation (ventral striatum + ventral medial prefrontal cortex) systems. With increased activity in reward-related brain regions, self-affirmation has been shown in multiple studies to influence stress-related physiological responses in both laboratory and real-life settings. For example, SA significantly reduce cortisol response to laboratory stress tasks, moderated by dispositional self-resources an indicator of hypothalamic-pituitary-adrenal (HPA) axis activity, with effects further influenced by dispositional self-resources. Studies have also been conducted to show a positive buffer effect of SA test on cardiovascular outcomes. For instance, one study revealed that SA tasks attenuate cardiovascular reactivity during negative emotion induction, as evidenced by lower maximum heart rate, higher respiratory sinus arrhythmia (RSA), and overall reduced ratings of negative affect.

Besides blood pressure and heart rate, one key measurement in this experiment is respiratory sinus arrhythmia (RSA). RSA is a form of heart rate variability and is defined as the variation between heart beats coincident with respiration. It is measured by calculating the R-R intervals (time between the R peaks) in the ECG waveform. RSA is controlled by the parasympathetic nervous system and has been shown to be an indicator of stress in laboratory settings. In this study, the investigators propose to measure participants' reactions to grieving stress by RSA. Consider participants' respiration pattern may be affected by sudden mood change during the grief recall task, the study team would also collect impedance cardiography data and use the measurement of respiration rate if needed. Impedance cardiography also provides measures of hemodynamic cardiovascular functioning such as cardiac output and total peripheral resistance.

While SA has been suggested to mitigate grief, its effect on grief has yet to be studied within laboratory settings. Previous studies have argued that "loss of self" is common among divorcing couples, who experience a loss that often involves grieving. Higher ratings of judge-rated loss of self are associated with higher endorsements of complicated grief symptoms among divorced couples. Given the potential for self-affirmation to enhance self-confidence and self-worth, it may also mitigate grief-related stress and physiological stress responses.

Study Protocol

Participants will be recruited from the SONA undergraduate participation pool of University of South Florida. Two RAs will be present during the lab visit. The primary RA is responsible for obtaining consent, guiding the experiment process, and conducting grief-recall interview. The secondary RA is responsible for collecting physiological data by operating the computer in the lab common area. The investigators will add RAs to the protocol through a MOD submitted the IRB.

The informed consent electronic document will be provided to the subjects as they arrive to the lab. After informed consent has been acquired, the subjects will be asked to complete several questionnaires including the Health Questionnaire, the Pre-task Grief Questionnaire, the Beck Depression Inventory (BDI), the Self-Worth Questionnaire (SWQ), the General Anxiety Disorder-7 (GAD-7), the Penn State Worry Questionnaire (PSWQ), the Pittsburgh Sleep Quality Index (PSQI), the Posttraumatic Stress Disorder Checklist (PCL-5), the Perceived Stress Scale (PSS-10), the Inclusion of Others in the Self Scale, the Global Meaning Violation Scale, the Social Relationships Index (SRI) and the Prolonged Grief Disorder (PG-13-Revised) Scale.

Next the participants' heights and weights will be measured, after which cardiovascular measurement equipment will be attached. Then, the participants will sit quietly as they watch an emotionally neutral nature video of Alaska. This rest period will last for 10 minutes, during which ECG impedance cardiography and blood pressure will be measured.

Once resting recordings are obtained, participants will be randomly assigned to the self-affirmation (SA) task or control tasks. The self-affirmation/control task will be administered for10 minutes, during which the study team will collect ECG, impedance cardiography and blood pressure measures. After the task, the subjects will complete self-worth questionnaire (SWQ) before the primary RA enters the room to perform the grief recall (GR) interview. The GR usually will be administered for 10 minutes, during which the study team will collect ECG, impedance cardiography and blood pressure measures.

Once the GR interview is finished, participants will be left alone in the room and instructed to sit quietly for 10 minutes for a recovery period. ECG, impedance cardiography and blood pressure measures will be taken throughout. After recovery, participants will finish the third part of questionnaires, including the third Self-Worth Questionnaire (SWQ), Grief Recall Response Questionnaire, Post-Grief Interview Questionnaire, and the Brief State Rumination Inventory. The research assistant will then conclude the study, thank, and compensate the participant.

Key Methods

Grief Recall: During the Grief Recall interview the PI will conduct a guided interview to promote feelings of grief in bereaved participants. The interview takes roughly ten minutes, during which research assistants ask participants to first recall a situation that happened after they experienced their loss and to wish their lost one was there with them. The grief recall interview has been shown to efficiently promote feelings of grief and elevate blood pressure in laboratory settings. Participants' grief severity was also found to be positively associated with their blood pressure reactivity, highlighting its relevance as a method for assessing cardiovascular outcomes. The GR interview was developed by one of our collaborators, Dr.Mary-Frances O'Connor. Dr. O'Connor has informed us that she has used grief recall in a number of studies with bereaved participants without any adverse events. She will also train the PI and study staff in administering the GR interview. Dr.O'Connor's affiliation to the study will be limited only to train the study PI and the study team. Dr.O'Connor will not be involve in the study procedures or any study activities. The study team do not intend to share identifiable information with Dr.O'Connor or any other collaborators unless permissions are obtained from our respective IRBs.

Self-affirmation intervention: Participants will be randomly assigned to either a self-affirming task or a non-affirming neutral task prior to engaging in grief recall. During the ten-minute self-affirmation task, participants will be asked to rank 11 values they may find important in their lives, and write about their top-ranked feature. This method has been shown to promote participant's self-awareness of their value and self-worth. Participants in no-affirmation control group will be asked to rank their top 12 favorite jellybean flavors and write about the 3rd and 4th favorite flavor for the same duration of time. This control task has also been tested to propose same amount of workload without promoting participants' self-worth.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 and older who have experienced the death of family member and/or friend within the last 2 to 18 months.
* Participants must also be fluent in English as all procedures will be conducted in English.

Exclusion Criteria:

- Individuals with a history of cardiovascular disease or disorders, those who report being pregnant, or are taking medication which may alter/affect cardiovascular and/or cognitive processes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Hypothesis 1: There will be a main effect of self-affirmation condition on CV reactivity and recovery to the grief recall task | Two months after the last participant data collection.
  A series of one-way ANCOVAs will be conducted to compare measures of cardiovascular reactivity and recovery between the self-affirmation and control conditions, controlling for gender, race, and baseline values, using a significance level of α = .05.
  CV reactivity will be operationalized as the difference between CV during grief recall and CV baseline measures.
  CV recovery will be operationalized as the difference between CV recovery measures and CV baseline measures.
Hypothesis 2: Grief severity (as measured by the PG-13 Questionnaire) will moderate the effect of the self-affirmation condition on cardiovascular reactivity and recovery. | Two months after the last participant.
  A series of multiple regression analyses will be conducted separately for HR, SBP, DBP and HF-HRV on reactivity and recovery. Predictor variables will include grief severity (PG-13 scores), experimental condition (value-affirmation vs. control, dummy-coded), and the condition x Grief Severity interaction. Dependent variables will be cardiovascular reactivity and recovery. A significant interaction would support the hypothesis that the effect of self-affirmation on reactivity and/or recovery is dependent on grief levels. It is predicted that the stress-buffering effect of self-affirmation will be strongest for individuals with high grief severity, evidenced by a smaller HR, SBP, and HF-HRV compared to the control group. The method calculating recovery would be the same as the method used in H1.
Hypothesis 3 (Exploratory): There will be a mediated moderation effect: the self-report measurement of self-worth mediates the change in cardiovascular reactivity, moderated by grief severity. | Two months after the last participant data collection.
  A moderated mediation analysis with Hayes PROCESS model will be conducted to explore whether the effect of value-affirmation on cardiovascular reactivity is mediated by changes in self-worth and moderated by grief severity. Change in self-worth will be operationalized by the difference in scores on the Self-Worth Questionnaire (SWQ) taken at timepoint 2 and 3 (right before and after the grief recall). The research team hypothesized that the self-worth variable will mediate the relationship between experimental condition and cardiovascular reactivity, with the relationship between self-worth and reactivity moderated by the participant's level of grief severity.
Hypothesis 4-1: Grief is related to psychological stress among young adult grieving participants: depression | Two months after the last participant.
  To test the hypothesis that grief severity is positively associated with participant's level of depression, a bivariate correlation will be conducted. Grief severity, as measured by scores on the prolonged grief (PG-13) questionnaire, will serve as the predictor variable. PG-13 includes 13 questions with a minimum value of 13 and a maximum value of 65, while higher value indicates higher level of grief. The outcome variable will be the scores of the Beck Depression Inventory (BDI). The BDI scale includes 21 questions with a minimum value of 0 and a maximum value of 63, where higher value indicates higher levels of depression. The research team proposed that participants scoring higher on PG-13 would also score higher in BDI, indicating greater vulnerability to depression.
Hypothesis 4-2: Grief is related to psychological stress among young adult grieving participants: anxiety | Two months after the last participant.
  To test the hypothesis that grief severity is positively associated with participant's anxiety level, a bivariate correlation will be conducted. Grief severity, as measured by scores on the prolonged grief (PG-13) questionnaire, will serve as the predictor variable. PG-13 includes 13 questions with a minimum value of 13 and a maximum value of 65, while higher value indicates higher level of grief. The outcome variable will be the scores of the Generalized Anxiety Disorder-7 scale (GAD-7). The GAD-7 scale includes 7 questions with a minimum value of 0 and a maximum value of 21, where higher value indicates higher levels of anxiety. The research team proposed that participants scoring higher on PG-13 would also score higher in GAD-7, indicating greater vulnerability to anxiety.
Hypothesis 4-3: Grief is related to psychological stress among young adult grieving participants: worries | Two months after the last participant.
  To test the hypothesis that grief severity is positively associated with participant's worriness level, a bivariate correlation will be conducted. Grief severity, as measured by scores on the prolonged grief (PG-13) questionnaire, will serve as the predictor variable. PG-13 includes 13 questions with a minimum value of 13 and a maximum value of 65, while higher value indicates higher level of grief. The outcome variable will be the scores of the Penn State Worry Questionnaire (PSWQ). The PSWQ scale includes 16 questions with a minimum value of 16 and a maximum value of 80, where higher value indicates higher levels of worriness. The research team proposed that participants scoring higher on PG-13 would also score higher in PSWQ, indicating greater levels of worriness.
Hypothesis 4-4: Grief is related to psychological stress among young adult grieving participants: perceived stress | Two months after the last participant.
  To test the hypothesis that grief severity is positively associated with participant's sleep quality, a bivariate correlation will be conducted. Grief severity, as measured by scores on the prolonged grief (PG-13) questionnaire, will serve as the predictor variable. PG-13 includes 13 questions with a minimum value of 13 and a maximum value of 65, while higher value indicates higher level of grief. The outcome variable will be the scores of the Perceived Stress Scale (PSS-10). PSS-10 scale includes 10 questions with a minimum value of 0 and a maximum value of 40, where higher value indicates higher levels of daily stress experienced within the last month. The research team proposed that participants scoring higher on PG-13 would also score higher in PSS, indicating greater levels of perceived stress.
Hypothesis 4-5: Grief is related to psychological stress among young adult grieving participants: sleep quality | Two months after the last participant.
  To test the hypothesis that grief severity is positively associated with participant's sleep disturbance, a bivariate correlation will be conducted. Grief severity, as measured by scores on the Prolonged Grief (PG-13) questionnaire, will serve as the predictor variable. PG-13 includes 13 questions with a minimum value of 13 and a maximum value of 65, while higher value indicates higher level of grief. The outcome variable will be the scores of the Pittsburgh Sleep Quality Index (PSQI). PSQI includes a mixture of likert-scale questions and short-answer questions that is transferrable to scores, with a minimum value of 0 and a maximum value of 21, where higher value indicates worst sleeping quality. The research team proposed that participants scoring higher on PG-13 would also score higher in PSQI, indicating greater levels of sleep disturbance.
Hypothesis 4-6: Grief is related to psychological stress among young adult grieving participants: Post-traumatic Stress Disorder | Two months after the last participant.
  To test the hypothesis that grief severity is positively associated with participant's PTSD symptoms, a bivariate correlation will be conducted. Grief severity, as measured by scores on the Prolonged Grief (PG-13) questionnaire, will serve as the predictor variable. PG-13 includes 13 questions with a minimum value of 13 and a maximum value of 65, while higher value indicates higher level of grief. The outcome variable will be the scores of the PTSD Checklist for DSM-5 (PCL-5). PCL-5 includes 20 questions with a minimum value of 0 and a maximum value of 80, where higher value indicates higher PTSD symptoms. The research team proposed that participants scoring higher on PG-13 would also score higher in PCL-5, indicating greater levels PTSD symptoms.
Hypothesis 5-1 (exploratory): Grief Severity is associated with meaning violation | Two months after the last participant.
  To test the hypothesis that grief severity is associated with higher meaning violation, linear regression will be conducted. Grief severity, as measured by scores on the prolonged grief (PG-13) questionnaire, will serve as the predictor variable. PG-13 includes 13 questions with a minimum value of 13 and a maximum value of 65, while higher value indicates higher level of grief. The outcome variable will be the scores of the Global Meaning Violation Scale (GMVS). GMVS includes 13 questions with a minimum value of 0 and a maximum value of 78, where higher value indicates higher levels meaning violation brought by the death event. The research team proposed that participants scoring higher on PG-13 would also score higher on GMVS, indicating higher level of meaning violation.
Hypothesis 5-2 (exploratory): Grief Severity is associated with perceived inclusion | Two months after the last participant.
  To test the hypothesis that grief severity is associated with higher inclusion of others in one's self, a linear regression will be conducted. Grief severity, as measured by scores on the prolonged grief (PG-13) questionnaire, will serve as the predictor variable. PG-13 includes 13 questions with a minimum value of 13 and a maximum value of 65, while higher value indicates higher level of grief. The outcome variable will be the scores of the Inclusion of Others in the Self Scale (IOS). IOS includes 2 subscales, each with a minimum value of 0 and a maximum value of 7, where higher value indicates higher levels of inclusion of other person or other group members to the self.
Hypothesis 5-3 (exploratory): Grief Severity is associated with complicated relationship | Two months after the last participant.
  To test the hypothesis that grief severity is associated with complicated relationship, a linear regression will be conducted. Grief severity, as measured by scores on the prolonged grief (PG-13) questionnaire, will serve as the predictor variable. PG-13 includes 13 questions with a minimum value of 13 and a maximum value of 65, while higher value indicates higher level of grief. The outcome variable will be the scores of the Social Relationship Index (SRI). SRI includes short-answer questions and likert-scale selections, with a minimum value of 4 and a maximum value of 24, where higher value indicates more complicated relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Salomon, Ph.D, Study Director — University of South Florida; Kaiyuan Luo, BS, BA, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Psychology and Communication Sciences and Disorders Lab Building, Tampa, Florida, United States

REFERENCES:
- [Background] Marchetti, I., Mor, N., Chiorri, C., Koster, E.H.W. (2024). Brief State Rumination Inventory (BSRI). In: Medvedev, O.N., Krägeloh, C.U., Siegert, R.J., Singh, N.N. (eds) Handbook of Assessment in Mindfulness Research. Springer, Cham. https://doi.org/10.1007/978-3-030-77644-2_119-1
- [Background] Campo, R.A., Uchino, B.N., Holt-Lunstad, J., Vaughn, A.A., Reblin, M., & Smith, T.W. (2009). The Assessment of Positivity and Negativity in Social Networks: The Reliability and Validity of the Social Relationships Index. Journal of Community Psychology, 37, 471-486. DOI: 10.1002/jcop.20308
- [Background] Prigerson HG, Horowitz MJ, Jacobs SC, Parkes CM, Aslan M, Goodkin K, Raphael B, Marwit SJ, Wortman C, Neimeyer RA, Bonanno GA, Block SD, Kissane D, Boelen P, Maercker A, Litz BT, Johnson JG, First MB, Maciejewski PK. Prolonged grief disorder: Psychometric validation of criteria proposed for DSM-V and ICD-11. PLoS Med. 2009 Aug;6(8):e1000121. doi: 10.1371/journal.pmed.1000121. Epub 2009 Aug 4. PMID 19652695
- [Background] Park, C. L., Riley, K. E., George, L. S., Gutierrez, I. A., Hale, A. E., Cho, D., & Braun, T. D. (2016). Global Meaning Violation Scale (GMVS) [Database record]. APA PsycTests. https://doi.org/10.1037/t65154-000
- [Background] Aron, A., Aron, E. N., & Smollan, D. (1992). Inclusion of Other in the Self Scale and the structure of interpersonal closeness. Journal of Personality and Social Psychology, 63(4), 596-612. https://doi.org/10.1037/0022-3514.63.4.596
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Meyer TJ, Miller ML, Metzger RL, Borkovec TD. Development and validation of the Penn State Worry Questionnaire. Behav Res Ther. 1990;28(6):487-95. doi: 10.1016/0005-7967(90)90135-6. PMID 2076086
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Tiwari R, Kumar R, Malik S, Raj T, Kumar P. Analysis of Heart Rate Variability and Implication of Different Factors on Heart Rate Variability. Curr Cardiol Rev. 2021;17(5):e160721189770. doi: 10.2174/1573403X16999201231203854. PMID 33390146
- [Background] Szuhany KL, Malgaroli M, Miron CD, Simon NM. Prolonged Grief Disorder: Course, Diagnosis, Assessment, and Treatment. Focus (Am Psychiatr Publ). 2021 Jun;19(2):161-172. doi: 10.1176/appi.focus.20200052. Epub 2021 Jun 17. PMID 34690579
- [Background] Sakuragi S, Sugiyama Y, Takeuchi K. Effects of laughing and weeping on mood and heart rate variability. J Physiol Anthropol Appl Human Sci. 2002 May;21(3):159-65. doi: 10.2114/jpa.21.159. PMID 12148458
- [Background] Saavedra Perez HC, Direk N, Milic J, Ikram MA, Hofman A, Tiemeier H. The Impact of Complicated Grief on Diurnal Cortisol Levels Two Years After Loss: A Population-Based Study. Psychosom Med. 2017 May;79(4):426-433. doi: 10.1097/PSY.0000000000000422. PMID 27879552
- [Background] Kim HG, Cheon EJ, Bai DS, Lee YH, Koo BH. Stress and Heart Rate Variability: A Meta-Analysis and Review of the Literature. Psychiatry Investig. 2018 Mar;15(3):235-245. doi: 10.30773/pi.2017.08.17. Epub 2018 Feb 28. PMID 29486547
- [Background] Fagundes CP, Wu EL. Matters of the heart: Grief, morbidity, and mortality. Curr Dir Psychol Sci. 2020 Jun 1;29(3):235-241. doi: 10.1177/0963721420917698. Epub 2020 May 7. PMID 33758475
- [Background] Critcher CR, Dunning D. Self-affirmations provide a broader perspective on self-threat. Pers Soc Psychol Bull. 2015 Jan;41(1):3-18. doi: 10.1177/0146167214554956. Epub 2014 Oct 15. PMID 25319717
- [Background] Creswell JD, Welch WT, Taylor SE, Sherman DK, Gruenewald TL, Mann T. Affirmation of personal values buffers neuroendocrine and psychological stress responses. Psychol Sci. 2005 Nov;16(11):846-51. doi: 10.1111/j.1467-9280.2005.01624.x. PMID 16262767
- [Background] Chen WJ, Nelson AM, Johnson HB, Fleming R. Effects of self-affirmation on emotion and cardiovascular responses. Stress Health. 2021 Apr;37(2):201-212. doi: 10.1002/smi.2986. Epub 2020 Sep 24. PMID 32954655
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Cascio CN, O'Donnell MB, Tinney FJ, Lieberman MD, Taylor SE, Strecher VJ, Falk EB. Self-affirmation activates brain systems associated with self-related processing and reward and is reinforced by future orientation. Soc Cogn Affect Neurosci. 2016 Apr;11(4):621-9. doi: 10.1093/scan/nsv136. Epub 2015 Nov 5. PMID 26541373
- [Background] Buckley T, Stannard A, Bartrop R, McKinley S, Ward C, Mihailidou AS, Morel-Kopp MC, Spinaze M, Tofler G. Effect of early bereavement on heart rate and heart rate variability. Am J Cardiol. 2012 Nov 1;110(9):1378-83. doi: 10.1016/j.amjcard.2012.06.045. Epub 2012 Jul 30. PMID 22853984
- [Result] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369